CLINICAL TRIAL: NCT02227537
Title: Evaluation of the Providence Nighttime Brace for the Treatment of Adolescence Idiopathic Scoliosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: OrthoGeorgia (Other)
Responsible Party: Principal Investigator, William Dasher, MD, Orthopaedic Spine Surgeon, OrthoGeorgia
Other Study IDs: OG12-04-13
Record Dates: First submitted 2014-08-22; First posted 2014-08-28 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Adolescence Idiopathic Scoliosis
Keywords: Adolescence Idiopathic Scoliosis; nighttime Bracing; Providence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adolescence idiopathic scoliosis: Patients must be at least 10 years of age with a risser score of 0, 1, or 2
  Interventions: Device: Providence Nighttime Bracing System

INTERVENTIONS:
Device: Providence Nighttime Bracing System — Providence Nighttime Bracing System
Device: Providence Nighttime Bracing System — The Providence brace is a polypropylene plastic, acrylic framed, system designed to apply corrective forces to scoliatic curves achieving correction or reduction of scoliosis.

SUMMARY:
A multicenter, prospective, non-randomized, single-arm observational study evaluating the Providence nighttime bracing system in patients diagnosed with adolescence idiopathic scoliosis.

DETAILED DESCRIPTION:
This study is designed as a multicenter, prospective, non-randomized, single arm observational study. A temperature probe and data logger will be attached to the Providence brace to monitor patient compliance wear time. Subjects will be blinded to temperature sensor readings to maximize objectivity of brace wear.

ELIGIBILITY:
Inclusion Criteria:

* Subject/guardian is able to provide informed consent and must sign the Institutional Review Board approved Informed Consent Form;
* Clinical/radiographic diagnosis of adolescence idiopathic scoliosis;
* Male/female;
* Skeletally immature (Risser grade 0, 1, or 2);
* Cobb angle between 25-40 degrees;
* Pre-menarchal or post-menarchal by no more than 1 year at the time of diagnosis;
* Curve apex caudal to T6 vertebrae;
* Physical and mental ability to adhere to bracing protocol;
* Have agreed to refuse participation in another clinical trial for the duration of the study.

Exclusion Criteria:

* History of previous surgical intervention or other invasive treatment for AIS;
* History of orthotic treatment or other brace wear for the treatment of AIS;
* Diagnosis of other musculoskeletal or developmental illness that might be responsible for the spinal curvature;
* Tumor or malignant tumor in the spine;
* Inability to communicate clearly in the English language;
* Subjects with a Risser score ≥ 3;
* Plans to relocate within the next 2 years;
* Any subject the Principle Investigator deems as an unfit candidate.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: up to 100 adolescent male/female will be enrolled at up to 4 sites in the US. Patients must be at least 10 years of age. Participants who receive treatment must have been diagnosed with adolescent idiopathic scoliosis without other significant spinal pathology. Appropriate participant selection will be accomplished through the integration of clinical and radiological parameters while ruling out other confounding sources of back pain or curvature. Subjects will be included who demonstrate a Cobb angle between 25-40 degrees. Participants must have radiographic evidence of a Risser grade of 0, 1, or 2. All chronic disease process and other possible sources for spinal curvature will be excluded by thorough history and physical examination.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Curve progression | subjects will be followed up for a period of 24 months from their first visit after receiving the Providence nighttime bracing system
  * The percentage of patients who have ≤5o curve progression and the percentage of patients who have ≥6 o progression at maturity;
  * The percentage of patients with curves exceeding 45o at maturity and the percentage who have had surgery recommended/undergone;
  * 2 year follow-up beyond maturity to determine the percentage of patients who subsequently undergo surgery.
  Routine follow-up visits will be scheduled 6 months apart (1st visit after brace fitting, 6, 12, 18 and 24 months) up to 24 months. At each of these visits, the patient will undergo a history & physical, PA radiographs, Cobb Angle assessment, Adams Forward Bending test, Neurological examination, outcome questionnaire's, concomitant medications, and adverse event recordings.

SECONDARY OUTCOMES:
Compliance | subjects will be followed up for a period of 24 months from their first visit after receiving the Providence nighttime bracing system
  A temperature data logger will record and monitor patient compliance of brace wear. To not create undue awareness to these recordings patients will be informed the temperature readings are being monitored for patient comfort and ease of brace wear. Reconciliation of data logger recordings will be conducted every 3 months.
Functionality | subjects will be followed up for a period of 24 months from their first visit after receiving the Providence nighttime bracing system
  Both study subjects and their guardians will be asked to fill out an Adolescent Health Assessment. Based on the Version 2.0 Pediatrics-Parent/ Adolescent Outcomes Instrument also commonly referred to as the PODCI ("Pediatric Outcomes Data Collection Instrument")
physical health and personal image | subjects will be followed up for a period of 24 months from their first visit after receiving the Providence nighttime bracing system
  Both study subjects and their guardians will be asked to fill out an Adolescent Health Assessment. Based on the Version 2.0 Pediatrics-Parent/ Adolescent Outcomes Instrument also commonly referred to as the PODCI ("Pediatric Outcomes Data Collection Instrument")

CONTACTS AND LOCATIONS:
Overall Officials: William B Dasher, MD, Principal Investigator — OrthoGeorgia; Eric D Lincoln, DO, Principal Investigator — Georgia Pediatric Orthopaedics; Winston R Jeshuran, MD, Principal Investigator — OrthoGeorgia; Wayne Kelley, MD, Principal Investigator — OrthoGeorgia; Randolph Devereaux, PhD, Principal Investigator — Mercer University School of Medicine; Hamza H Awad, MD, PhD, Principal Investigator — Mercer University School of Medicine
Locations (2):
- United States (2):
  - Georgia Pediatric Orthopaedics, Macon, Georgia
  - OrthoGeorgia, Macon, Georgia